CLINICAL TRIAL: NCT02506348
Title: Comparison of Diclofenac vs. Nepafenac Ophthalmic Drops: Patient Comfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Asaf Achiron, Dr.Asaf Achiron, Wolfson Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: 0011-15
Record Dates: First submitted 2015-07-02; First posted 2015-07-23 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Post Surgical Management; Pain Management; Inflamation Management
MeSH Terms: conditions — Agnosia | interventions — Diclofenac; nepafenac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diclofenac+Nepafenac (Experimental): one drop Diclofenac in one eye one drop Nepafenac in other eye
  Interventions: Drug: Diclofenac; Drug: Nepafenac

INTERVENTIONS:
Drug: Diclofenac
Drug: Nepafenac

SUMMARY:
In this study we test Diclofenac and Nepafenac and compared patients experience and comfort following administration of these ophthalmic drops.

DETAILED DESCRIPTION:
In this study we will compare the ocular tolerability between preservative-free Diclofenac and Nepafenac drops. Using a standard comparative scale we will measured discomfort, itching, burning and pain in intervals of 1 sec, 5 sec, 1 min and 5 min post-administration.

The results may aid both doctors and patients in decision regarding the post surgical anti-inflammatory treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient facing cataract surgery

Exclusion Criteria:

* under 18
* cognitive decline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
patient's comfort | 1 min post administration
  change in patient's comfort between both eyes at 1 min post administration

SECONDARY OUTCOMES:
patient's comfort | 5 min post administration
  change in patient's comfort between both eyes at 10 min post administration

CONTACTS AND LOCATIONS:
Locations (1):
- The E.Wolfson Medical Center, Holon, Israel